CLINICAL TRIAL: NCT00193375
Title: Phase II Trial of Concurrent Irinotecan, Carboplatin and Radiation Therapy Followed by Bevacizumab (Avastin) in the Treatment of Patients With Limited Stage Small Cell Lung Cancer
Brief Title: Irinotecan, Carboplatin and Radiation Therapy Followed by Bevacizumab in Limited Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry); Pharmacia and Upjohn (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 72
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2012-11-13 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Irinotecan; Carboplatin; Bevacizumab; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Patients received carboplatin [area under the concentration-versus-time curve of 5 intravenously (IV) day 1 every 3 weeks x 4), irinotecan (50mg/m2 IV days 1 and 8 every 3 weeks x 4], and radiation (1.8 Gy daily to a total of 61.2 Gy beginning with the 3rd cycle). Cycles 3 and 4 were 28 days each; with restaging after 4 cycles. Patients without progressive disease received bevacizumab (10 mg/kg IV every 14 days x 10).
  Interventions: Drug: Irinotecan; Drug: Carboplatin; Drug: Bevacizumab; Radiation: Radiation

INTERVENTIONS:
Drug: Irinotecan — 50mg/m2 days 1 & 8 each 21-day cycle 1 & 2, 28-day cycle 3 & 4
  Other Names: Camptosar
Drug: Carboplatin — AUC 5
  Other Names: Paraplatin
Drug: Bevacizumab — 10mg/kg IV every 2 weeks for 10 doses starting week 16
  Other Names: Avastin
Radiation: Radiation

SUMMARY:
In this multicenter trial, we plan to evaluate the feasibility and toxicity of initial treatment with irinotecan/carboplatin/radiation therapy, followed by treatment with bevacizumab, in patients with limited stage small cell lung cancer.

DETAILED DESCRIPTION:
Upon determination of eligibility, all patients will be receive:

* Irinotecan + Carboplatin + Radiation Therapy + Bevacizumab

Patients will receive 4 courses of irinotecan/carboplatin. Radiation therapy will begin concurrently with the third course of chemotherapy. The intervals between chemotherapy courses will be 21 days except for the interval between the third and fourth courses (during radiation therapy), which will be 28 days.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Small cell lung cancer, confirmed by biopsy.
* Limited stage disease after standard evaluation.
* Able to perform activities of daily living without assistance.
* No previous treatment with chemotherapy, radiation therapy, or biologics.
* Measurable or evaluable disease
* Adequate bone marrow, liver and kidney function
* Able to understand the nature of this study and give written consent.

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Age < 18 years
* History of previous malignancies
* Women pregnant or lactating
* History or physical exam evidence of central nervous system disease)
* Active infection requiring intravenous antibiotics
* Full-dose anticoagulation or thrombolytic therapy within 10 days
* Proteinuria.
* Serious nonhealing wound, ulcer, or bone fracture
* Evidence if bleeding diathesis or coagulopathy
* History of heart attack within 6 months.
* Uncontrolled cardiovascular disease
* PEG or G-tube
* History of other serious disease

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-08; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC

REFERENCES:
- [Background] Spigel DR, Greco FA, Zubkus JD, Murphy PB, Saez RA, Farley C, Yardley DA, Burris HA 3rd, Hainsworth JD. Phase II trial of irinotecan, carboplatin, and bevacizumab in the treatment of patients with extensive-stage small-cell lung cancer. J Thorac Oncol. 2009 Dec;4(12):1555-60. doi: 10.1097/JTO.0b013e3181bbc540. PMID 19875975

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 60
Completed | 41
Not Completed | 19

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: years] | 65 [42 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Secondary Outcome: 2-Year Progression-free Survival (PFS)
Description: Progression-free survival (PFS) was defined as the date of study entry until the date of tumor progression or death. 2-Year PFS is the percentage of patients alive and without progressive disease (PD) 2 years from the date of study entry.
Time Frame: 24 months
Population: All patients were assessed for progression free survival.
Measure: Number; unit: percentage of participants
Arm/Group | Intervention
Number analyzed (Participants) | 60
percentage of participants | 22

2. Secondary Outcome: Overall Response Rate
Description: Overall response rate is the percentage of patients with complete response or partial response per RECIST v.1 Criteria. Complete response (CR) = Disappearance of all target lesions, disappearance of all nontarget lesions for at least 4 weeks. Partial Response (PR) = At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameters.
Time Frame: 18 month
Population: All patients were evaluated for response by RECIST v. 1 criteria. All patients with major responses had confirmation of response on repeat scans by the same technique(s) 4 weeks (or longer) later.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intervention
Number analyzed (Participants) | 60
percentage of participants | 80 [68 to 89]

3. Primary Outcome: Number of Grade 3/4 Toxicities Patients Experienced on Maintenance Bevacizumab Following Chemoradiation for Limited Stage - Small Cell Lung Cancer (LS-SCLC)
Description: Toxicity was evaluated in all patients who received at least 1 dose of therapy, and graded according to CTCAE v. 3.
Time Frame: 18 months
Population: Patients who received at least one dose of bevacizumab maintenance therapy were assessed for toxicities.
Measure: Number; unit: Grade 3/4 Toxicity Events
Arm/Group | Intervention
Number analyzed (Participants) | 41
Grade 3/4 Toxicity Events
  Hemorrhage | 2
  Diarrhea | 1
  Fatigue | 1
  Hypertension | 1
  Nausea | 1
  Infection - Other (Pnemonia) | 4
  Pulmonary toxicities | 4
  Leukopenia | 2
  Neutropenia | 1
  Thrombocytopenia | 1

ADVERSE EVENTS:
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 35/60
Other Adverse Events (participants affected / at risk) | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=60)
Pulmonary/Upper Respiratory - Other (Acute respiratory failure) (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhage, GI (Upper GI NOS) (Blood and lymphatic system disorders) | 2
Infection - Other (Aspergillus pneumonia) (Infections and infestations) | 1
Dehydration (Gastrointestinal disorders) | 1
Death not associated with CTCAE term (Disease Progression NOS) (General disorders) | 3
Fistula, GI - esophagus (Gastrointestinal disorders) | 1
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1
Infection - Other (influenza) (Infections and infestations) | 1
Infection with Grade 3/4 Neutrophils - Blood (Infections and infestations) | 1
Infection - Other (obstructive pneumonia) (Infections and infestations) | 1
Perforation, GI - Colon (Gastrointestinal disorders) | 1
Infection with unknown ANC - Lung (pnemonia) (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 6
Thrombosis/thrombus/embolism (Vascular disorders) | 4
Pulmonary fibrosis (radiographic changes) (Respiratory, thoracic and mediastinal disorders) | 1
Seizure (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=60)
Alopecia (Skin and subcutaneous tissue disorders) | 4
Neutrophils (Blood and lymphatic system disorders) | 53
Anorexia (Gastrointestinal disorders) | 22
Mood Alteration - Anxiety (Psychiatric disorders) | 4
Pain - joint (General disorders) | 3
Pain - back (General disorders) | 3
Constipation (Gastrointestinal disorders) | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dehydration (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 28
Dizziness (Nervous system disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 5
Edema (General disorders) | 8
Esophagitis (Gastrointestinal disorders) | 9
Fatigue (General disorders) | 51
Hemorrhage, Pulmonary/upper respiratory (Blood and lymphatic system disorders) | 6
Hemoglobin (Blood and lymphatic system disorders) | 57
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 3
Infection (Infections and infestations) | 3
Insomnia (General disorders) | 3
Pain - muscle (Musculoskeletal and connective tissue disorders) | 3
Nausea (Gastrointestinal disorders) | 44
Platelets (Blood and lymphatic system disorders) | 55
Pulmonary Symptoms (Respiratory, thoracic and mediastinal disorders) | 24
Rash (Skin and subcutaneous tissue disorders) | 16
Vomiting (Gastrointestinal disorders) | 21
Leukocytes (Blood and lymphatic system disorders) | 56
Fatigue (General disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.